CLINICAL TRIAL: NCT03240419
Title: Probiotic Supplementation in Obese Pregnant Women. A Feasibility Study.
Brief Title: Prenatal Probiotic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 203392
Record Dates: First submitted 2017-07-24; First posted 2017-08-07 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Childhood Obesity; Maternal Obesity During Childbirth; Insulin Resistance; Inflammation
Keywords: Obesity; Inflammation; Pregnancy; Programming
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance; Inflammation; Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Each probiotic capsule contains 180 mg of a standardized white to light beige fine powder consisting of freeze-dried cultures. Specifically, Bifidobacterium BB-12® and Lactobacillus rhamnosus LGG® (50%:50%). This product has a minimum potency of 6.5 billion (6.5E+9) CFU (ColonyForming Units) per capsule. Other ingredients in the powder are: microcrystalline cellulose, maltodextrin, silicon dioxide and magnesium stearate. Participants in this group will take one daily capsule orally starting at the time of recruitment (gestation week 12) and until delivery.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Participants in this group will take one capsule containing microcrystalline cellulose, maltodextrin, silicon dioxide and magnesium stearate (all ingredients listed in the probiotic capsules except the culture) . Participants in this group will take one daily capsule orally starting at the time of recruitment (gestation week 12) and until delivery.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Bifidobacterium BB12 and Lactobacillus Rhamosus LGG (50%:50%) capsules.
  Other Names: live cultures
  Arms: Probiotics
Dietary Supplement: Placebo — capsule manufactured to mimic probiotic capsules.
  Arms: Placebo

SUMMARY:
This study will assess the feasibility of a randomized control trial in which the effects of probiotic supplementation throughout pregnancy on maternal insulin sensitivity and inflammation, as well offspring gene expression and body composition are examined.

DETAILED DESCRIPTION:
Maternal obesity leads to increased insulin resistance and inflammation which have been shown to induce fetal adaptations and greater risk of obesity in the offspring. Probiotic supplementation during pregnancy has been shown to improve insulin sensitivity in normal weight women. However, little is known on the effects of probiotic supplementation throughout pregnancy on maternal insulin sensitivity and inflammation as well as offspring gene expression and body composition. Long term nutritional supplementation, however, is associated with increased participant burden as well as lower compliance and retention rates. Thus, this study will assess the feasibility of a long term probiotic supplementation study in obese pregnant women. Acceptance and compliance with daily capsules throughout pregnancy and study procedures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30
* ≥ 18 years of age
* Singleton pregnancy
* Less than 12 weeks of gestation
* Less than 1 serving of yoghurt with live cultures or cultured milk per week
* Conceived without assisted fertility treatments

Exclusion Criteria:

* • Women with pre-existing medical conditions (e.g., diabetes, hypertension, thyroid disorders, heart disease or immune disorders) as determined by the PI to affect the outcomes of interest

  * Immunosuppressed women
  * Women taking medications during pregnancy known to affect fetal growth (i.e., thyroid hormone, glucocorticoids, insulin, oral hypoglycemic agents)
  * Women who are using recreational drugs, tobacco or alcohol during their pregnancy
  * Milk intolerance or allergy
  * Consuming probiotic supplements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is on pregnant women.
Enrollment: 60 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Change in acceptance of probiotic supplementation throughout pregnancy in obese women. | Self-administered questionnaires will be done at gestation weeks 12,14, 18, 22, 26, 30 and 36
  Participants will answer acceptability questionnaires in which they will have to rate (1= poor, 2= fair, 3= good, 4= very good, and 5= excellent ) their experience with capsule supplementation and study procedures.
Change in compliance with probiotic supplementation throughout pregnancy in obese women. | Pill count will be done at gestation weeks 12,14, 18, 22, 26, 30 and 36
  Change in compliance with capsule supplementation will be assessed during pregnancy via pill-count.

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Diaz Fuentes, MD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

REFERENCES:
- [Background] Allen SJ, Jordan S, Storey M, Thornton CA, Gravenor M, Garaiova I, Plummer SF, Wang D, Morgan G. Dietary supplementation with lactobacilli and bifidobacteria is well tolerated and not associated with adverse events during late pregnancy and early infancy. J Nutr. 2010 Mar;140(3):483-8. doi: 10.3945/jn.109.117093. Epub 2010 Jan 20. PMID 20089774
- [Background] Dugoua JJ, Machado M, Zhu X, Chen X, Koren G, Einarson TR. Probiotic safety in pregnancy: a systematic review and meta-analysis of randomized controlled trials of Lactobacillus, Bifidobacterium, and Saccharomyces spp. J Obstet Gynaecol Can. 2009 Jun;31(6):542-552. doi: 10.1016/S1701-2163(16)34218-9. PMID 19646321
- [Background] Ilmonen J, Isolauri E, Poussa T, Laitinen K. Impact of dietary counselling and probiotic intervention on maternal anthropometric measurements during and after pregnancy: a randomized placebo-controlled trial. Clin Nutr. 2011 Apr;30(2):156-64. doi: 10.1016/j.clnu.2010.09.009. PMID 20970896
- See also: Arkansas Children's Nutrition Center website — https://acnc.uams.edu/home/studies/